CLINICAL TRIAL: NCT06003894
Title: Comparison of the Effectiveness of Kegel Exercises and 360-degree Expanded Diaphragm Breathing Pattern Training in Individuals With Urinary Incontinence
Brief Title: 360 Degree Expanded Diaphragm Breathing Pattern Training in Individuals With Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Dr. Öğr. Üyesi Ömer Şevgin, Asst. Prof. Dr., Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Uskudar64
Record Dates: First submitted 2023-08-15; First posted 2023-08-22 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Urinary Incontinence
Keywords: kegel exercises; urinary incontinence; diaphragmatic breathing
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Intervention Model Description: 360 degree expanded diaphragm breathing
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- kegel group (Active Comparator): Participants will only practice kegel exercises.
  Interventions: Other: kegel exercises
- diaphragm group (Experimental): In addition to kegel exercises, 360 degree expanded diaphragm breathing training will be given to the participants.
  Interventions: Other: kegel exercises; Other: 360 degree expanded diaphragmatic breathing training

INTERVENTIONS:
Other: kegel exercises — Kegel exercises; It is done by squeezing your pelvic floor muscles for 3 to 5 seconds and relaxing them. Participants are expected to do this exercise in the form of hold-relax 10-15 times each set. Participants are expected to practice Kegel exercises, 2 sets a day, 3 days a week for 8 weeks.
Other: 360 degree expanded diaphragmatic breathing training — 360-degree expanded diaphragm breathing is the delivery of air taken during inspiration to the postero-lateral wall of the abdomen. Breathing in this way ensures that the pressure in the abdomen is distributed equally in all directions. Practices for using this breathing pattern will be done 2 sets per day, each set for 10 minutes.
  Arms: diaphragm group

SUMMARY:
The aim of this study is to investigate the effect of transferring the healthy intra-abdominal pressure created by 360 degree expanded diaphragm breathing taught to the patient to the pelvic cavity on incontinence problems.

DETAILED DESCRIPTION:
66 people with a score of 3 or higher on the Incontinence Severity Index will be included in the study. All participants will complete the King Health Questionnaire and Incontinence Quality of Life Questionnaires. The control group will consist of 33 people and will apply only Kegel exercises 2 sets a day, 3 days a week for 8 weeks. The experimental group will consist of 33 people and the participants will apply Kegel exercises for 8 weeks, 3 days a week, 2 sets a day. In addition to this, 360 degree expanded diaphragm breathing training will be given to the experimental group. Practices for using this breathing pattern will be done 2 sets per day, each set for 10 minutes. At the end of 8 weeks, all 3 questionnaires will be asked to be filled again. The variation between the initial results and the final results, as well as the differences between the final changes, will also be compared.

ELIGIBILITY:
Inclusion Criteria:

* Getting a score of 3 and above in the incontinence severity index.
* Be in the age range of 12-65 years.
* No neurological problems.

Exclusion Criteria:

• Having a history of surgery or childbirth in the last 3 months.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2023-12-10 (Actual)

PRIMARY OUTCOMES:
The incontinence severity index (ISI) | 10 weeks
  It was developed in epidemiological and clinical studies to identify women with urinary incontinence of varying severity. The questionnaire score is obtained by multiplying the value given to the frequency of urinary incontinence by the value given to the amount of urinary incontinence. The result obtained; classified as mild, moderate, severe, very severe.
Understanding King's Health Questionnaire (KHQ) | 10 weeks
  The King's Health questionnaire is a two-part questionnaire that includes 32 items and is frequently used to evaluate the quality of life of patients with incontinence. It includes 7 sub-headings consisting of multiple items in addition to two single-item questions such as general health status and impact on quality of life. These include: role limitations, physical limitations, social limitations, limitations in personal relationships, emotional problems, sleep and energy disturbances associated with incontinence, and severity measures for incontinence. The second part is the 11-item Symptom Severity Scale, which assesses the presence and severity of urinary symptoms. The score of the Symptom Severity Scale ranges from 0 (best) to 30 (worst). For other areas, scores range from 0 (best) to -100 (worst).
Incontinence Quality of Life Questionnaire (I-QOL) | 10 weeks
  In the Incontinence Quality of Life Scale (I-QOL), which consists of 22 items, all items are evaluated on a five-category Likert-type scale (1= a lot, 2= a lot, 3= moderately, 4= a little, 5= not at all). The scores of the questionnaire and its subscales are obtained by adding the scores of each item and dividing this total by the number of items. For easier explanation of the scores, the calculated total score is converted to a scale value from 0 (lowest quality of life) to 100 (highest quality of life). High scores indicate better quality of life than low scores.

CONTACTS AND LOCATIONS:
Overall Officials: Elif AKAR, Study Chair — Uskudar University
Locations (1):
- Üsküdar Unıversıty, Üsküdar, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang YC, Chang KV. Kegel Exercises. 2023 May 1. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK555898/ PMID 32310358
- [Background] Cho ST, Kim KH. Pelvic floor muscle exercise and training for coping with urinary incontinence. J Exerc Rehabil. 2021 Dec 27;17(6):379-387. doi: 10.12965/jer.2142666.333. eCollection 2021 Dec. PMID 35036386
- [Background] Singla N, Aggarwal H, Foster J, Alhalabi F, Lemack GE, Zimmern PE. Management of Urinary Incontinence Following Suburethral Sling Removal. J Urol. 2017 Sep;198(3):644-649. doi: 10.1016/j.juro.2017.02.3341. Epub 2017 Mar 4. PMID 28267602
- [Background] Snodgrass W, Barber T. Comparison of bladder outlet procedures without augmentation in children with neurogenic incontinence. J Urol. 2010 Oct;184(4 Suppl):1775-80. doi: 10.1016/j.juro.2010.04.017. Epub 2010 Aug 21. PMID 20728128
- [Background] Abu Raddaha AH, Nasr EH. Kegel Exercise Training Program among Women with Urinary Incontinence. Healthcare (Basel). 2022 Nov 24;10(12):2359. doi: 10.3390/healthcare10122359. PMID 36553882